CLINICAL TRIAL: NCT04284293
Title: Clinical Study to Assess Safety and Efficacy of Subretinal Injection of Human Neural Progenitor Cells for Treatment of Retinitis Pigmentosa
Brief Title: CNS10-NPC for the Treatment of RP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Clive Svendsen, Director, Regenerative Medicine Institute, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Study00000375
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Retinitis Pigmentosa
Keywords: RP; Retinopathy; Pigmentary Retinopathy; Retinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1A (Experimental): Visual acuity of 20/200 or worse
  Single, unilateral, subretinal injection of 300,000 CNS10-NPC (n=3)
  Interventions: Biological: CNS10-NPC implantation
- Group 1B (Experimental): Visual acuity of 20/200 or worse
  Single, unilateral, subretinal injection of 1,000,000 CNS10-NPC (n=3)
  Interventions: Biological: CNS10-NPC implantation
- Group 2 (Experimental): Visual acuity between 20/80 and 20/200
  Single, unilateral, subretinal injection of 1,000,000 CNS10-NPC (n=10)
  Interventions: Biological: CNS10-NPC implantation

INTERVENTIONS:
Biological: CNS10-NPC implantation — All patients will receive a single, unilateral, subretinal injection of CNS10-NPC
  Other Names: Neural Progenitor Cell (NPC); Stem Cell

SUMMARY:
The investigator is examining the safety of transplanting cells into the subretinal space of patients with Retinitis Pigmentosa (RP). The cells are called neural progenitor cells, which are a type of stem cell that can become several different types of cells in the nervous system. These cells have been derived to specifically become astrocytes, which is a type of neuronal cell. The cells are called "CNS10-NPC." The investigational treatment has been tested in animals, but it has not yet been tested in people. In this study, the investigators want to learn if CNS10-NPC cells are safe to transplant into the subretinal space of people.

DETAILED DESCRIPTION:
This study will be the first to use a human progenitor cell line to treat retinitis pigmentosa in people. This is a Phase 1/2a, single-center, open label, safety study of two escalating doses of human neural progenitor cells (CNS10-NPC) delivered unilaterally to the subretinal space of subjects with RP.

Subjects meeting all Eligibility Criteria and providing Informed Consent will be enrolled in one of two sequential dosing groups. Subjects will be treated sequentially with a minimum of one month interval between surgeries for the first three subjects in each dosing cohort. The remaining subjects in the cohort will be treated with a minimum interval of at least one week between surgeries.

Primary objective. To assess the safety and tolerability of two escalating doses of clinical grade human fetal cortical-derived neural progenitor cells (CNS10-NPC) administered in the subretinal space of one eye (unilaterally) in patients with retinitis pigmentosa (RP).

Secondary objectives. Within constraints of a small first in-human study focused on safety:

1. Determine if CNS10-NPC can engraft and survive long-term in the retina of transiently immunosuppressed subjects,
2. Obtain evidence that subretinal injection of CNS10-NPC can favorably impact the progression of vision loss in subjects with moderate RP.

ELIGIBILITY:
Inclusion Criteria:

1. To participate in this study, the subject must be 18 years of age or older and must understand and sign the protocol's informed consent.
2. Participant with diagnosis of retinitis pigmentosa.

   * Clinical signs of retinitis pigmentosa.
   * A history of nyctalopia
   * Retinal pigmentary changes
   * Arteriolar attenuation
   * Waxy disc pallor
   * Electrophysiologic evidence of rod dysfunction on full field electroretinography
   * Visual field constriction.

     3a. Participants in Group 1 (n=6) will have visual acuity equal to or worse than 20/200. Participants in Group 2 (n=10) will have visual acuity equal to or worse than 20/80.

     3b. Group 1 participants will have central visual field of 40 degrees diameter or less. Group 2, participants will have a measurable visual field defect.

4. Participant will be medically able to undergo ophthalmic surgery.

Exclusion Criteria:

1. Presence of significant ocular abnormalities that would preclude the planned surgery or interfere with the interpretation of study endpoints (e.g. glaucoma, corneal or significant lens opacities, pre-existing uveitis, intraocular infection, macular edema, choroidal neovascularization). Any ocular diseases that the investigator feels would interfere with accurate ocular measurements. This would exclude potential subjects with significant cataract, corneal scars or significant corneal irregularities such as keratoconus, previous penetrating keratoplasty or glaucoma with central visual field.
2. Any pre-existing factor or history of eye disease that may predispose to an increased risk of surgical complications in the study eye (e.g. trauma, previous surgery other than uncomplicated cataract surgery, uveitis, congenital developmental or structural abnormalities).
3. Concomitant systemic diseases including those in which the disease itself, or the treatment for the disease, can alter ocular function or immune status (e.g. malignancies, uncontrolled diabetes).
4. Any ocular surgery or laser in either eye within 12 weeks of screening.
5. Any contraindication to pupil dilatation in either eye.
6. Treatment with intravitreal, subtenon or periocular steroid within 4 months of enrollment.
7. Any known allergy to any component of the delivery vehicle or diagnostic agents used during the study (e.g., dilation drops), or medications planned for use during the peri-operative period including corticosteroids, tacrolimus and mycophenolate.
8. Imminently life-threatening illness.
9. Abuse of alcohol or any illegal substance(s) within 12 months of the procedure.
10. Laboratory test abnormalities or abnormalities in electrocardiogram or chest X-ray, which in the opinion of the Principal Investigator are clinically significant and would make the patient unable to tolerate study procedures.
11. Intercurrent illness or infection 28 days prior to enrolment.
12. Contraindications to use of anesthesia.
13. Females of child-bearing potential (i.e. those who are not surgically sterile and not at least 12-months post-menopausal) who are not willing to comply with the study's contraception requirement (women who are unwilling to use an effective form of contraception such as the contraceptive pill or intrauterine device).
14. Women who are pregnant.
15. Females who are nursing or who intend to nurse during the first 6 months post-treatment.
16. Men or women who do not agree to use barrier or medical contraception for at least 6 months post-operatively.
17. History of any investigational agent administration within 28 days prior to administration.
18. Participation in a prior gene transfer therapy study or cell-based therapy.
19. Enrollment in any other clinical study, for any condition, including those relating to RP throughout the duration of the study.
20. Current or anticipated long-term treatment with systemic corticosteroids (for a period longer than 7 days).
21. Current treatment with immunosuppressant therapies or any contraindications to use of the immunosuppressants in this protocol.
22. A history of malignancy within a five-year period or a positive cancer screening test within a one-year period of the screening visit.
23. Any physical or mental disability that will impair the ability of the patient to travel to and from the study center or provide informed consent/assent or effective safety assessments as specified by the protocol. Any mental or psychiatric disorders that prevent the patient from having full authority to do so (i.e. the subject cannot have power of attorney signed over to another individual).
24. Inability or unwillingness to comply with the study protocol.
25. Medical history of HIV, or hepatitis A, B or C.
26. Subjects who have taken any prescription or investigational oral retinoid medication (e.g., Accutane® Soriatane®), or any medicines that may affect the macula (e.g. tamoxifen, mellaril, thorazine, plaquenil, niacin) within 6 months of enrollment.
27. Allergy to Beta-Lactam antibiotics.
28. The presence of cystoid macular edema.
29. Glucose-6-phosphate dehydrogenase (G6PD) Deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety as evaluated by incidence of Adverse Events (AE) and Serious Adverse Events (SAE) and their relationship to the intervention | Subjects will be followed postoperatively for 12 months
Safety, as evaluated by changes in the complete blood count | Subjects will be followed postoperatively for 12 months
Safety, as evaluated by changes in the comprehensive metabolic panel | Subjects will be followed postoperatively for 12 months
Safety, as evaluated by changes in Donor Specific Antibodies | Subjects will be followed postoperatively for 12 months
Safety, as evaluated by changes in the urinalysis | Subjects will be followed postoperatively for 12 months
Safety, as evaluated by changes in Visual Acuity | Subjects will be followed postoperatively for 12 months
  ETRDS, or FrACT in cases of very low vision.
Safety, as evaluated by changes in visual field | Subjects will be followed postoperatively for 12 months
  Goldman perimetry will be used for central visual fields and microperimetry will be used for peripheral visual fields
Safety, as evaluated by changes in Spectral Domain Optical Coherence Tomography (SD-OCT) | Subjects will be followed postoperatively for 12 months
  Ellipsoid zone measurement through SD-OCT will be performed

SECONDARY OUTCOMES:
Slit lamp examination | Performed 7 times over 15 months
Intraocular pressure measurement | Performed 7 times over 15 months
Funduscopic examination | Performed 7 times over 15 months
Fundus photography (color, red free, or infrared) | Performed 4 times over 15 months
Fundus Autofluorescence (FAF) | Performed 4 times over 15 months
Best Corrected Visual Acuity | Performed 7 times over 15 months
Visual Function Questionnaire-25 (VFQ-25) | Performed 5 times over 15 months
  The Visual Function Questionnaire-25 is graded in a scale from 0-100 where a higher number represents better function
Spectral domain optical coherence tomography (SD-OCT) | Performed 5 times over 15 months
  Retinal Thickness
Electroretinography (ERG) | Performed 5 times over 15 months
Goldmann visual field area (microperimetry) | Performed 5 times over 15 months
Change in rate of vision field loss | Through study completion, ~15 months.

CONTACTS AND LOCATIONS:
Overall Officials: David Liao, MD, PhD, Principal Investigator — Retina-Vitreous Associates Medical Group
Locations (1):
- Retina-Vitreous Associates Medical Group, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu B, Avalos P, Svendsen S, Zhang C, Nocito L, Jones MK, Pieplow C, Saylor J, Ghiam S, Block A, Fernandez M, Ljubimov AV, Small K, Liao D, Svendsen CN, Wang S. GMP-grade human neural progenitors delivered subretinally protect vision in rat model of retinal degeneration and survive in minipigs. J Transl Med. 2023 Sep 25;21(1):650. doi: 10.1186/s12967-023-04501-z. PMID 37743503